CLINICAL TRIAL: NCT04572646
Title: Benefit of a Systematic Proposition of Nicotine Replacement Therapy Preoperatively for Patients Undergoing Planned Surgery and With Tobacco or Cannabis Addiction, Regardless of the Intention to Quit
Brief Title: Benefit of Systematic Proposition of Nicotine Substitution for Patients Undergoing Surgery
Acronym: PATCHIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment goal not feasible
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020/03-ECR-GHMG
Record Dates: First submitted 2020-09-15; First posted 2020-10-01 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-03

CONDITIONS: Smoking Cessation
Keywords: postoperative complication; nicotine replacement therapy; exhaled carbon monoxide level
MeSH Terms: conditions — Smoking Cessation; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NRT proposition and exhaled CO measurement (Other)
  Interventions: Other: NRT proposition and exhaled CO measurement

INTERVENTIONS:
Other: NRT proposition and exhaled CO measurement — Nicotine replacement therapy is proposed to every patient included in the study.
  Whether the patient accepts the therapy or not, exhaled carbon monoxide is measured at the preoperative consultation (about 15 days before surgery) and the day of surgery by a nurse. These two measures are compared to assess efficacy of nicotine replacement therapy.

SUMMARY:
Smoking is associated with a higher rate of surgical complications. For example, in orthopedics, the risk of complications is 31% in smokers against 5% in non-smokers. The management of this addiction is recommended and particularly interesting in scheduled surgery, because it allows smoking cessation well before the procedure. However, for patients who cannot consider this smoking cessation, the mere information of the risk cannot be sufficient and a real strategy must be constructed and evaluated.

Currently, studies results indicate that a patient reducing the number of smoked cigarettes will unconsciously modify their smoking behaviour to obtain the usual nicotine level, this effect is called self-titration. Conversely, nicotine replacement while continuing consumption could induce an improvement in smoking behaviour, therefore less intoxication which would be beneficial in terms of reduction of post-operative complications. This study seeks to assess the effectiveness of a systematic proposition of nicotine replacement therapy (NRT) in regular smokers. Tobacco addiction specialists have demonstrated that intoxication and dependence are well correlated with the exhaled carbon monoxide (CO) level, so this measurement will be used in addition to the patient's interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient who smokes at least one cigarette or cannabis joint per day, every day
* Patient received for nurse consultation at least 48 hours before surgery
* Patient planned to undergo surgery, with entry the day of surgery and 1 day of post-operative hospitalisation
* Patient in physical capacity and willing to undergo exhaled carbon monoxide measurement
* For patients with one of the following chronic diseases: diabetes, Chronic Obstructive Pulmonary Disease, glucose intolerance, hemolytic anemia, asthma and dilation of the bronchi, these diseases must be stable
* Signature of the specific study informed consent
* Patient affiliated or beneficiary of social security system

Exclusion Criteria:

* Inability to submit to study follow-up for geographic, social or psychological reasons
* Patient already included in an interventional clinical research protocol
* Patients protected by French law from clinical research inclusion (pregnant, in labour, breastfeeding, legally protected, under judiciary or administrative liberty deprivation)
* Patient using nicotine substitutes before the nurse consultation
* Alcohol consumption six hours before the exhaled carbon monoxide measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of a systematic proposition of nicotine replacement therapy, regardless of the intention to quit Change in exhaled carbon monoxide level between the two measurements, assessed by a carbon monoxide breath monitor | At inclusion, and before surgery

SECONDARY OUTCOMES:
Number of patients who refuse nicotine replacement therapy | At inclusion
Effect of nicotine replacement therapy on the type of analgesics administrated | At inclusion, before surgery, and 2 days after surgery
Effect of nicotine replacement therapy on the duration of analgesics administrated | At inclusion, before surgery, and 2 days after surgery
Effect of nicotine replacement therapy on the dose of analgesics administrated | At inclusion, before surgery, and 2 days after surgery
Number of smoking cessations | 2 days after surgery
Efficacy of a systematic proposition of nicotine replacement therapy, depending on the intention to quit Change in exhaled carbon monoxide level between the two measurements, assessed by a carbon monoxide breath monitor | At inclusion, and before surgery
  Subgroup analysis of the primary endpoint according to predefined groups

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Mutualiste de Grenoble, Grenoble, France